CLINICAL TRIAL: NCT00118573
Title: Randomized Clinical Trial Comparing Surveillance and Selective Surgical Treatment for Abdominal Aortic Aneurysms Less Than 5.5 cm in Diameter Versus Early Endovascular Treatment
Brief Title: Comparison of Surveillance Versus Aortic Endografting for Small Aneurysm Repair
Acronym: CAESAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lower than anticipated events;slow recruitment;larger than predicted sample size
Sponsor: University Of Perugia (Other)
Collaborators: William Cook Europe (Industry)
Responsible Party: Principal Investigator, Piergiorgio Cao, MD, Professor of Vascular Surgery, University Of Perugia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 384/03
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Aortic Aneurysm, Abdominal; Endovascular
Keywords: abdominal aortic aneurysm; randomized controlled trial; endovascular aneurysm repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVAR (Experimental): AAA repair with endografting
  Interventions: Procedure: EVAR (Endovascular repair of Abdominal Aortic aneurysm)
- Surveillance (Active Comparator): Not AAA repair; surveillance
  Interventions: Procedure: Surveillance

INTERVENTIONS:
Procedure: EVAR (Endovascular repair of Abdominal Aortic aneurysm) — AAA repair with endografting
  Other Names: early endovascular repair of abdominal aortic aneurysm; repair of abdominal aneurysm by aortic endografting
  Arms: EVAR
Procedure: Surveillance — Surveillance of AAA without any repair until AAA will reach 5.5cm, become tender or rapidly grow
  Other Names: monitoring abdominal aortic aneurysm without repair
  Arms: Surveillance

SUMMARY:
Objective of the present study is to compare endovascular repair versus surveillance and, eventually delay treatment in patients with small abdominal aortic aneurysms (AAA), with respect to patient survival, AAA rupture and AAA related death risks.

DETAILED DESCRIPTION:
The study will include patients with small AAA (diameter 4.1 to 5.4 cm defined by Computed Tomographic scan) suitable for endovascular repair (EVAR).

Randomization is designed with equal probability of assignment to each of the two groups (ie, immediate endovascular repair or surveillance group) by means of a computer-generated -random-number list . After eligibility is verified, assignment will be made using a computer database held at the Coordinating Centre.

In the immediate repair group, endovascular repair with introduction of an aortic endograft (Cook Zenith) will be performed within six weeks from randomization.

In the surveillance group, patients are followed without repair until the aneurysm reaches 5.5 cm in diameter, or enlarges at least 1.0 cm in one year, or until patient develops symptoms that are attributed to the aneurysm by the attending investigator. When one of these criteria is met, endovascular repair (if the patient remains a candidate for EVAR), or open repair will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 50-80 years of age
* Non symptomatic infrarenal AAA of 4.1 to 5.4 cm in diameter measured by CT performed within 3 months before randomization
* Adequate infrarenal aortic neck (length > 15 mm diameter < 30 mm) and other anatomical configurations suitable for EVAR
* Patients have a life expectancy of at least 5 years
* Signed informed consent

Exclusion Criteria:

* Ruptured or symptomatic AAA
* AAA maximum diameter >= 5.5 cm
* Suprarenal or thoracic aorta aneurysm of more than 4.0 cm
* Patient unsuitable for administration of contrast agent
* Severe heart, lung, liver or renal disease (serum creatinine >= 3mg/dl)
* Need for adjunctive major surgical or vascular procedures within 1 month
* High likelihood of non compliance with follow-up requirements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2004-09; Primary Completion 2010-05 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
all cause mortality at 3 years | 3 years

SECONDARY OUTCOMES:
aneurysm related mortality at 3 years | 3 years
aneurysm rupture rates at 3 years | 3 years
perioperative or late complications | 30 days and 3 years
conversion to open repair | 30 days and 3 years
loss of treatment options | 3 years
risks associated with delayed treatment | 30 days and 3 years
aneurysm growth rates | 3 years
quality of life | 30 days, 6 month, 1 year, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Piergiorgio Cao, MD, Principal Investigator — University Of Perugia
Locations (20):
- Vitkovice Hospital Ostrava and University Hospital Ostrava - Poruba, Ostrava, Czechia
- Hopital Cardiologique CHRU, Lille, France
- Germany (2):
  - University of Koeln, Cologne
  - Klinik Fuer Gefasschirurgie st.Franziskus Hospital, Münster
- Carmel Medical Center, Haifa, Israel
- Italy (9):
  - U.O.Chirurgia Vascolare Az Osp Carrara, Carrara
  - Dip Chirurgia Vascolare Osp S.Anna, Ferrara
  - Chirurgia Vascolare Az Osp Careggi, Florence
  - Chirurgia Vascolare Ospedale San Giovanni di Dio, Florence
  - Chirurgia Vascolare, Ospedale San Donato, Milan
  - Azienda Ospedaliera "Antonio Cardarelli", Napoli
  - S.C. Chirurgia Vascolare - Università di Perugia, Perugia
  - S.C. Chirurgia Vascolare Az Osp. S.Maria Nuova, Reggio Emilia
  - Policlinico Le Scotte - U.O. Chirurgia Vascolare, Siena
- Catharina Ziekenhuis, Eindhoven, Netherlands
- Poland (2):
  - Klinika Chirurgii ogolnej i Chorob Klatki Piersiowej Warsaw, Warsaw
  - Naczyniowej i Transplantacyjnej Akademii Medycznej, Warsaw
- Spain (2):
  - Institute of Cardiovascular Disease Hospital Clinic University of Barcelona, Barcelona
  - Complejo Hospitalario, Toledo
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- [Background] Alcorn HG, Wolfson SK Jr, Sutton-Tyrrell K, Kuller LH, O'Leary D. Risk factors for abdominal aortic aneurysms in older adults enrolled in The Cardiovascular Health Study. Arterioscler Thromb Vasc Biol. 1996 Aug;16(8):963-70. doi: 10.1161/01.atv.16.8.963. PMID 8696960
- [Background] Scott RA, Wilson NM, Ashton HA, Kay DN. Is surgery necessary for abdominal aortic aneurysm less than 6 cm in diameter? Lancet. 1993 Dec 4;342(8884):1395-6. doi: 10.1016/0140-6736(93)92756-j. PMID 7901685
- [Background] United Kingdom Small Aneurysm Trial Participants; Powell JT, Brady AR, Brown LC, Fowkes FG, Greenhalgh RM, Ruckley CV, Thompson SG. Long-term outcomes of immediate repair compared with surveillance of small abdominal aortic aneurysms. N Engl J Med. 2002 May 9;346(19):1445-52. doi: 10.1056/NEJMoa013527. PMID 12000814
- [Background] Mortality results for randomised controlled trial of early elective surgery or ultrasonographic surveillance for small abdominal aortic aneurysms. The UK Small Aneurysm Trial Participants. Lancet. 1998 Nov 21;352(9141):1649-55. PMID 9853436
- [Background] Lederle FA, Wilson SE, Johnson GR, Reinke DB, Littooy FN, Acher CW, Ballard DJ, Messina LM, Gordon IL, Chute EP, Krupski WC, Busuttil SJ, Barone GW, Sparks S, Graham LM, Rapp JH, Makaroun MS, Moneta GL, Cambria RA, Makhoul RG, Eton D, Ansel HJ, Freischlag JA, Bandyk D; Aneurysm Detection and Management Veterans Affairs Cooperative Study Group. Immediate repair compared with surveillance of small abdominal aortic aneurysms. N Engl J Med. 2002 May 9;346(19):1437-44. doi: 10.1056/NEJMoa012573. PMID 12000813
- [Background] EVAR trial participants. Endovascular aneurysm repair versus open repair in patients with abdominal aortic aneurysm (EVAR trial 1): randomised controlled trial. Lancet. 2005 Jun 25-Jul 1;365(9478):2179-86. doi: 10.1016/S0140-6736(05)66627-5. PMID 15978925
- [Derived] De Rango P, Verzini F, Parlani G, Cieri E, Romano L, Loschi D, Cao P; Comparison of surveillance vs. Aortic Endografting for Small Aneurysm Repair (CAESAR) Investigators. Quality of life in patients with small abdominal aortic aneurysm: the effect of early endovascular repair versus surveillance in the CAESAR trial. Eur J Vasc Endovasc Surg. 2011 Mar;41(3):324-31. doi: 10.1016/j.ejvs.2010.11.005. Epub 2010 Dec 9. PMID 21145269
- [Derived] Cao P, De Rango P, Verzini F, Parlani G, Romano L, Cieri E; CAESAR Trial Group. Comparison of surveillance versus aortic endografting for small aneurysm repair (CAESAR): results from a randomised trial. Eur J Vasc Endovasc Surg. 2011 Jan;41(1):13-25. doi: 10.1016/j.ejvs.2010.08.026. Epub 2010 Sep 25. PMID 20869890